CLINICAL TRIAL: NCT02313727
Title: Combined Treatment With TNF (Tumor Necrosis Factor) Inhibitor and Pamidronate in AS Patients: Effect on the Radiographic Progression
Brief Title: Combined Treatment With TNF Inhibitor and Pamidronate in AS Patients: Effect on the Radiographic Progression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0099-14-BNZ
Record Dates: First submitted 2014-12-01; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-11

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Pamidronate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pamidronate (Active Comparator): pamidronate
  Interventions: Drug: Pamidronate
- placebo (Placebo Comparator): placebo
  Interventions: Other: Placebo (NaCl 0.9%)

INTERVENTIONS:
Drug: Pamidronate — intravenous infusion of pamidronate 60 mg
  Arms: pamidronate
Other: Placebo (NaCl 0.9%) — intravenous infusion of NaCl 0.9% 500 ml
  Arms: placebo

SUMMARY:
It will be a pilot, 2 year, prospective, randomized, double-blind, placebo-controlled (for pamidronate) study. All patients with AS will receive treatment with TNF inhibitor, while randomization will be performed for pamidronate versus placebo group. Primary outcome will be the rate of radiographic progression of AS, calculated after 24 months of combined treatment.

DETAILED DESCRIPTION:
It will be a pilot, 2 year, prospective, randomized, double-blind, placebo-controlled (for pamidronate) study. All patients with AS will receive treatment with tumor necrosis factor (TNF) inhibitor, as indicated by local guidelines. Randomization will be performed for pamidronate vs placebo group. Pamidronate will be prescribed as monthly intravenous infusion in the dose of 60 mg/month for the first 6 consecutive months of every study year. Primary outcome will be the rate of radiographic progression of ankylosing spondylitis (AS), calculated after 24 months of combined treatment. Clinical and laboratory disease parameters will serve as secondary outcomes. These outcomes as well as safety assessments will be performed on a monthly basis up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* presence of spinal syndesmophytes
* normal renal and liver function
* eligibility to receive anti-TNF treatment according to local guidelines

Exclusion Criteria:

* unwilling to sigh the informed consent
* presence of significant systemic or organ-limited disorders, other than AS
* any contraindication for anti-TNF or pamidronate treatment
* presence of acute dental/periodontal disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
modified stock ankylosing spondylitis spine (mSASS) score | 24 months
  calculated by X-ray films of the spine
Bath ankylosing spondylitis radiographic index (BASRI) | 24 months
  calculated by X-ray films of the spine

SECONDARY OUTCOMES:
Bath ankylosing spondylitis disease activity index (BASDAI) | monthly from the date of randomization up to 24 months
  calculated
Ankylosing spondylitis disease activity index (ASDAS) | monthly from the date of randomization up to 24 months
  calculated
Bath ankylosing spondylitis functional index (BASFI) | monthly from the date of randomization up to 24 months
  calculated
Bath ankylosing spondylitis metrology index (BASMI) | monthly from the date of randomization up to 24 months
  calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

REFERENCES:
- [Background] Slobodin G, Rosner I, Feld J, Rimar D, Rozenbaum M, Boulman N, Odeh M. Pamidronate treatment in rheumatology practice: a comprehensive review. Clin Rheumatol. 2009 Dec;28(12):1359-64. doi: 10.1007/s10067-009-1256-2. Epub 2009 Aug 19. PMID 19690938
- [Background] Slobodin G, Rosner I, Rimar D, Boulman N, Rozenbaum M, Odeh M. The synergistic efficacy of adalimumab and pamidronate in a patient with ankylosing spondylitis. Clin Rheumatol. 2010 Jul;29(7):793-4. doi: 10.1007/s10067-010-1378-6. Epub 2010 Jan 29. PMID 20111975
- [Background] Pederson L, Ruan M, Westendorf JJ, Khosla S, Oursler MJ. Regulation of bone formation by osteoclasts involves Wnt/BMP signaling and the chemokine sphingosine-1-phosphate. Proc Natl Acad Sci U S A. 2008 Dec 30;105(52):20764-9. doi: 10.1073/pnas.0805133106. Epub 2008 Dec 15. PMID 19075223